CLINICAL TRIAL: NCT00947193
Title: A Phase 2a Study of Ataluren (PTC124) as an Oral Treatment for Nonsense-Mutation-Mediated Hemophilia A and B
Brief Title: Study of Ataluren (PTC124) in Hemophilia A and B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to Sponsor decision and not reflective of adverse safety findings.
Sponsor: PTC Therapeutics (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-011-HEM
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia A; Hemophilia B; Factor VIII; Factor IX; FVIII; FIX; Nonsense mutation; Premature stop codon; HA; HB; PTC124; Ataluren
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren Overall Study (Experimental): Ataluren was provided as a vanilla-flavored powder to be mixed with water or milk. Ataluren was taken 3 times per day, with dosing based on the participant's body weight. The dose level for ataluren was 5 mg/kg in the morning, 5 mg/kg at midday, and 10 mg/kg in the evening or 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 14 days, followed by an interval of 14 days without treatment.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Oral powder
  Other Names: PTC124

SUMMARY:
Hemophilia A (HA) and hemophilia B (HB) are inherited bleeding disorders caused by mutations in the gene for factor VIII (FVIII) and factor IX (FIX), respectively. These proteins are essential for blood clotting. The lack of FVIII/FIX can produce bleeding episodes that cause damage of the bone, muscles, joints, and tissues. A specific type of mutation, called a nonsense (premature stop codon) mutation, is the cause of the disease in approximately 10-30% of participants with hemophilia and results in severe manifestations. Ataluren (PTC124) is an orally delivered, investigational drug that acts to overcome the effects of the premature stop codon, potentially enabling the production of functional FVIII/FIX. This study is a Phase 2a trial evaluating the safety and efficacy of ataluren in participants with HA or HB due to a nonsense mutation. The main purpose of this study is to understand whether ataluren can safely increase FVIII/FIX activity levels.

DETAILED DESCRIPTION:
In this study, participants with hemophilia A or hemophilia B due to a nonsense mutation were treated with an investigational drug called ataluren (PTC124). Evaluation procedures to determine if a participant qualifies for the study was performed within 14 days prior to the start of treatment. Eligible participants who elected to enroll in the study then participated in a 28-day treatment period. Within the 28-day period, ataluren (PTC124) treatment was to be taken for 2 cycles of 14 days each 3 times per day with meals at a dose level of 5, 5, 10 milligrams/kilograms (mg/kg) in the first cycle and a dose level of 20, 20, 40 mg/kg in the second cycle. After the first 14-day cycle, study doses were changed to 10 mg/kg (morning), 10 mg/kg (midday), and 20 mg/kg (evening) and the doses were administered for 1 cycle only. Then, there was an interval of approximately 14 days without treatment. During the study, ataluren (PTC124) efficacy, safety, and pharmacokinetics were evaluated periodically with measurement of FVIII/FIX activity and inhibitor levels, other blood tests, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age ≥18 years
* Presence of a nonsense mutation as the sole disease-causing mutation in the FVIII or FIX gene
* At least 20 prior treatments with FVIII or FIX concentrates
* Willingness and ability to comply with scheduled visits, drug administration plan, study restrictions, and study procedures

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug
* Any history of prior anti-FVIII/FIX inhibitors
* Unable or unwilling to forego prophylactic FVIII/FIX concentrate use during the screening and on-study periods (Note: Participants were allowed use of FVIII/FIX concentrates for treatment of bleeding episodes while on study)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10-14 (Actual); Primary Completion 2011-08-30 (Actual); Study Completion 2011-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Barth, MD, Principal Investigator — PTC Therapeutics
Locations (13):
- United States (7):
  - The Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - New England Hemophilia Center, Worcester, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Hemostatis and Thrombosis Clinic, Nashville, Tennessee
  - Puget Sound Blood Center, Seattle, Washington
- St. Paul's Hospital, Vancouver, British Columbia, Canada
- France (3):
  - Hôpital Cardiologique, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Necker Enfants Malades, Paris
- Italy (2):
  - Azienda Ospedaliero-Universitaria Careggi Viale G.B. Morgagni, Florence
  - A.Bianchi Bonomi Hemophilia and Thrombosis Center, Milan

REFERENCES:
- [Background] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- [Background] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- See also: PTC Therapeutics' website — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, participants with HA or HB due to a nonsense mutation were recruited for the study.
Pre-assignment Details: Participants requiring treatment with Factor 8 (FVIII)/Factor 9 (FIX) concentrate during 14-day ataluren treatment could continue ataluren treatment for at least 14 days following discontinuing FVIII concentrate treatment for hemophilia type A (HA) and for at least 18 days following discontinuing FIX concentrate treatment for hemophilia type B (HB)
Groups:
- 5 mg/kg, 5 mg/kg, and 10 mg/kg Ataluren: Ataluren was provided as a vanilla-flavored powder to be mixed with water or milk. Ataluren was taken 3 times per day, with dosing based on the participant's body weight. The dose level for ataluren was 5 milligrams/kilograms (mg/kg) in the morning, 5 mg/kg at midday, and 10 mg/kg in the evening for 14 days, followed by an interval of 14 days without treatment.
- 10 mg/kg, 10 mg/kg, and 20 mg/kg Ataluren: Ataluren was provided as a vanilla-flavored powder to be mixed with water or milk. Ataluren was taken 3 times per day, with dosing based on the participant's body weight. The dose level for ataluren was 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 14 days, followed by an interval of 14 days without treatment.
Period: Overall Study
Arm/Group | 5 mg/kg, 5 mg/kg, and 10 mg/kg Ataluren | 10 mg/kg, 10 mg/kg, and 20 mg/kg Ataluren
Started | 3 | 10
Received at Least 1 Dose of Study Drug | 3 | 10
Completed | 0 | 10
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Factor VIII >1% | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Arm/Group | Ataluren Overall Study
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Plasma FVIII/FIX Activity Response at Day 14
Description: A plasma FVIII/FIX activity response was defined as an end-of-treatment (Day 14) activity of ≥1%.
Time Frame: Baseline up to Day 14
Population: All enrolled participants who received at least 1 dose of study drug and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg, 10 mg/kg, and 20 mg/kg Ataluren
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Number of Participants With a Change From Baseline in Plasma Anti-FVIII/FIX Inhibitor Titers at Day 14
Description: To assess the change from Baseline in plasma anti-FVIII/FIX inhibitor titers, it was determined if any potential antibodies were neutralizing using the Bethesda assay. The Bethesda assay demonstrates antibodies that are neutralizing by quantifying residual FVIII/FIX activity in normal plasma after serial dilutions with participant plasma. For this assay, the neutralizing antibody threshold value was 0.6 Bethesda units (BU).
Time Frame: Baseline and Day 14
Population: All enrolled participants who received at least 1 dose of study drug and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg, 10 mg/kg, and 20 mg/kg Ataluren
Number analyzed (Participants) | 10
Participants | 1

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs) by Severity and Relationship to Study Drug
Description: The relationship of TEAEs and SAEs to the study drugs was assessed as: probable related, possible related, unlikely related, and unrelated. The severity of TEAEs were graded using the Common Terminology Criteria for Adverse Events, Version 3.0, as: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening), or Grade 5 (fatal). A summary of other non-serious adverse events (AEs) and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Day 28
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren Overall Study
Number analyzed (Participants) | 13
Participants
  TEAEs | 8
  TEAEs Related to Study Drug | 2
  Severe TEAEs | 0
  SAEs | 0

4. Secondary Outcome: Number of Participants With a Clinically Meaningful Abnormal Clinical Laboratory (Hematology, Adrenal Assays, Biochemistry, and Urinalysis) Parameters
Description: The Investigator used his/her judgment in determining whether an abnormality was clinically significant, diagnostic evaluation was warranted, and potential interruption of ataluren was appropriate. Life-threatening (Grade 4) or severe (Grade 3) laboratory abnormalities were considered dose-limiting, although recurrent or persistent moderate (Grade 2) events were also considered dose-limiting in certain circumstances. Values considered abnormal included -Hematology: Serum total bilirubin Grade 2 (>1.5-3.0*upper limit of normal [ULN]) and Serum alanine aminotransferase, Serum aspartate aminotransferase, and Serum gamma glutamyl transferase Grade 2 (>2.5-3.0*ULN); -Adrenal: Plasma adrenocorticotropic hormone >ULN (and cortisol within normal limits); and -Renal: serum creatinine Grade 1 (>ULN-1.5*ULN) and Serum blood urea nitrogen ≥1.5-3.0*ULN. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Day 28
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable clinical laboratory data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren Overall Study
Number analyzed (Participants) | 13
Participants
  Hematology Assays: number analyzed (Participants) | 4
  Hematology Assays | 0
  Biochemistry Assays | 0
  Adrenal Assays | 0
  Urinalysis | 1

5. Secondary Outcome: Compliance With Ataluren Administration
Description: Ataluren compliance as assessed by quantification of used and unused drug. Data were not collected or analyzed for this measure because participants were terminated early from the study.
Time Frame: Baseline up to Day 28
Population: All enrolled participants who received at least 1 dose of study drug, completed the study, and had evaluable compliance with ataluren administration data.
Arm/Group | Ataluren Overall Study
Number analyzed (Participants) | 0

6. Secondary Outcome: Ataluren Plasma Exposure
Description: The ataluren plasma concentrations before and 2 hours after the first morning dose at end of treatment was measured.
Time Frame: Day 10 (pre-dose) and Day 14 (post-dose)
Population: All enrolled participants who received at least 1 dose of study drug, completed the study, and had evaluable plasma data.
Measure: Median (Full Range); unit: microgram/milliliters (μg/mL)
Arm/Group | 10 mg/kg, 10 mg/kg, and 20 mg/kg Ataluren
Number analyzed (Participants) | 10
microgram/milliliters (μg/mL)
  Pre-Dose: number analyzed (Participants) | 9
  Pre-Dose | 14.7 [5.94 to 28.7]
  Post-Dose: number analyzed (Participants) | 9
  Post-Dose | 6.66 [1.04 to 28.3]

7. Secondary Outcome: Occurrence of Bleeding Episodes
Description: Frequency, timing, anatomic location, and severity of any bleeding episodes were recorded. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 28
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren Overall Study
Number analyzed (Participants) | 13
Participants
  Participants Who Experienced a Bleeding Episode | 3
  Spontaneous Right Hip Bleed | 1
  Soft Tissue Bleed | 1
  Right Knee Bleed | 1
  Upper Shoulder Bleed | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: Adverse event data were collected from all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Ataluren Overall Study
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren Overall Study (N=13)
Diarrhoea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haemorrhage (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.